CLINICAL TRIAL: NCT04563364
Title: Interdisciplinary Hospital-home Intervention on the Adaptation of Motor Development in Premature Children.Randomized Clinical Trial
Brief Title: Interdisciplinary Hospital-home Intervention on Motor Development in Premature Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENF-32-2019
Record Dates: First submitted 2020-08-25; First posted 2020-09-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Premature Birth
Keywords: Infant; Child Development; Nursing; Physical Therapy Specialty
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospital-Home (Experimental): This group will receive an interdisciplinary intervention of education to parents for get better outcomes of motor development.
  Interventions: Other: Interdisciplinary hospital-home intervention
- Control Intervention (Active Comparator): Control group will receive a conventional treatment given by the institutions
  Interventions: Other: Convencional treatment

INTERVENTIONS:
Other: Interdisciplinary hospital-home intervention — The intervention will start in NICU and to be continued at home with the support of ICT. The NICU intervention will have theoretical and practical components, the theoretical one will be about motor development in premature infants, and practical one will have strategies for motor early intervention, it will be demonstrated with pediatric simulator and parents should be demonstrate it with a infant: 1Sensorial motor stimulation, visual and auditory follow-6up; Tactile integration 3Extension muscle activation 4Middle line integration 5Alignment reaction stimulation in prone position 6Flexor muscle activation with transition to lateral position 7Flexor muscle activation with transition to sitting position 8Facilitation of reciprocal flexion and extension lower limbs. All parents will receive a motor sensorial kit that will include roller, visual tags, blankets and rattles, it will be for apply the strategies for motor early intervention, and will be supported by ICT
  Arms: Hospital-Home
Other: Convencional treatment — Control group will receive a conventional treatment given by the institutions
  Arms: Control Intervention

SUMMARY:
Motor development of the premature infant often exhibits deviations that trigger functional limitations and disability. In Colombia, one out of every five births corresponds to premature babies. In preterm infants requiring hospitalization, early clinical interventions focused on home care have been shown to improve motor development and decrease morbidity.

However, interdisciplinary work, supported by information and communication Technologies (ICT), shows a knowledge gap that can be explored. This leads to the following research question: ¿What is the effect of an interdisciplinary Hospital-Home intervention addressing motor development adaptation in premature infants in Colombia in comparison with traditional interventions?

Objective: To determine the effect of an interdisciplinary Hospital-Home intervention addressing motor development adaptation in premature infants in Colombia in comparison with traditional interventions

Methodology Experimental quantitative study with pre-test and post-test to two groups, experimental and control, which compares before and after the intervention. The intervention will be developed in two scenarios: the hospital and the home. The experimental group will receive the intervention and the control group the traditional care established in the institutions for premature children. The calculation of the sample size is 130 participants.

Type of results expected to be obtained It is expected to obtain a supported that justifies the importance of education from hospital stay, post discharge follow-up and parental participation in the adequate stimulation of motor development of the premature. It is expected to incorporate the use of ICT in home monitoring, while implementing the use of a mobile application for this purpose. It is also expected to contribute to the research training of undergraduate and graduate students. In addition, participate in national and international presentations and in the production of scientific articles.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants between 34 and 37 weeks of gestation,
* Infants with weight over 1800gr
* Hemodynamic stability
* Interns in NICU of participants institutions (Colombia and Poland).
* Infants with residence in a places close to the institutional health care services.

Exclusion Criteria:

* Premature child with a musculoskeletal deformity.
* Premature child with diagnosis of a genetic syndrome
* Premature child with congenital heart diseases.
* Premature child with brain injuries.

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Motor Development. | 18 Months
  Test on infant motor performance (TIMPSI)

SECONDARY OUTCOMES:
CapDMP questionnaire | From enrollment to the end of treatment
  Questionnaire that measure the degree of knowledge in parents or caregivers about motor development in premature

CONTACTS AND LOCATIONS:
Overall Officials: Adriana L Castellanos, Mg., Principal Investigator — Universidad de la Sabana
Locations (1):
- Hospital San Rafael, Tunja, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandoval-Cuellar C, Castellanos-Garrido AL, Ospina Romero AM, Boude Figueredo OR, Serrano-Gomez ME, Fuya Caro CA, Molina Cardenas DC, Pinto Rosas EM. Motor development in premature infants: Study protocol for an interdisciplinary hospital-home intervention. Pediatr Neonatol. 2023 Sep;64(5):577-584. doi: 10.1016/j.pedneo.2022.12.015. Epub 2023 Mar 15. PMID 37002053